CLINICAL TRIAL: NCT07136233
Title: Evaluating the Impact of Educational Flyers Promoting $0 Deductibles and Lower Costs With Silver Plans on California Marketplace Plan Enrollment and Care Utilization
Brief Title: Impact of Benefit Inserts on Health Plan Selection and Utilization Among Renewing Covered California Members
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Covered California (Other Government)
Responsible Party: Principal Investigator, Sulo Paudyal, Research Data Specialist, Covered California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CCA-NOTICE-INSERT-2025
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Outreach Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Flyer Group (No Intervention): Renewing Covered California households who do not receive the informational flyer insert during the 2025 plan year. They only receive a standard renewal notice informing them of their upcoming coverage renewal and encourages consumers to shop for coverage ahead of the next coverage year.
- Flyer Group (Experimental): Renewing Covered California members who receive the informational flyer insert during the 2025 plan year along with a standard renewal notice informing them of their upcoming coverage renewal and encourages consumers to shop for coverage ahead of the next coverage year.
  Interventions: Behavioral: Informational Flyer Insert on Enhanced Silver Plan Benefits

INTERVENTIONS:
Behavioral: Informational Flyer Insert on Enhanced Silver Plan Benefits — Alongside the standard eligibility notice informing participants about their upcoming coverage renewal, an informational flyer is also included. The flyer explains that everyone is eligible in 2025 for the Silver plan regardless of income and highlights its benefits, such as $0 deductibles, lower monthly premiums, free preventive visits, and reduced costs for primary care, emergency care, and medications.
  Arms: Flyer Group

SUMMARY:
The study aims to evaluate the impact of an informational flyer insert on health plan selection and health care utilization among Covered California renewing members during the 2025 plan year. The flyer highlights the enhanced Silver plan benefits, which were expanded in 2025 to include all enrollees, regardless of income level. Key benefits include $0 deductibles, lower monthly premiums, free preventive visits, and reduced costs for primary care, emergency care, and medications.

The main questions the study seeks to answer are:

* Does the informational flyer help overcome barriers that prevent consumers from switching to more beneficial plans?
* Does the flyer encourage current Silver Plan enrollees to increase health care utilization, such as preventive visits, primary care, and medication usage, by highlighting enhanced benefits like $0 deductible and lower costs?

To address these questions, researchers will compare outcomes between households that receive the flyer insert and those that do not. Covered California's administrative data will provide individual-level information on plan selection, while claims data will offer insights into healthcare utilization patterns. This approach will help determine the effectiveness of targeted communication in driving selection of more beneficial plan and improving healthcare utilization.

DETAILED DESCRIPTION:
Background:

The Affordable Care Act (ACA) established health insurance marketplaces (commonly referred to as ACA marketplaces) to provide affordable insurance coverage. In addition to premium subsidies, administered through the form of advanced premium tax credits (APTCs), low-income consumers are eligible for reduced out-of-pocket costs when they enroll in a Silver plan through the ACA marketplaces. These ACA benefits, known as Cost-Sharing Reductions (CSRs), improve the plan generosity (through the form of lower copays and deductibles) while keeping premium costs at the level of a Silver plan. Traditionally, lower out-of-pocket costs are associated with higher premium payments, such as in the Platinum tier, whereas high out-of-pocket costs are paired with lower premiums, as in the Bronze tier. These CSR benefits are available for consumers who enroll in the Silver metal tier and have an income below 250 percent of the Federal Poverty Level (FPL).

California launched its own state-funded Cost-Sharing Reduction (CSR) program in 2024, increasing the benefit levels for those eligible for federally funded CSRs. These plans are referred to as "enhanced CSR plans." In the 2025 plan year, California expanded eligibility for enhanced CSR plans to all enrollees, regardless of income. This policy change improves affordability and accessibility by offering coverage comparable to Gold plans but with lower monthly premiums for all enrollees. Members already enrolled in Silver plans were automatically upgraded to the enhanced CSR plans, while those in other metal tiers (Bronze, Gold, or Platinum) had to take action to switch during the annual renewal period to benefit from these new plan designs. This study explores how additional communication in the form of an informational flyer insert about the new enhanced CSR plan benefits and their expanded eligibility may have helped overcome inertia, likely due to informational and awareness barriers, for renewing consumers.

Project Objective:

The primary objective of the study is to evaluate whether including an informational flyer insert with renewal notices affects consumer behavior in two key areas:

1. Enrollment in Enhanced CSR Plans: Assess whether members currently enrolled in other metal tiers are more likely to switch to the enhanced CSR plan when informed about the new benefits.
2. Health Care Utilization for Current Silver Plan Enrollees: Determine whether members already enrolled in Silver plans, who were newly eligible for enhanced silver benefits, increased their utilization of health care services after receiving the flyer insert which has information such as '$0 deductible', 'Lower monthly premiums', '$0 for preventative visits', 'lower costs for primary and emergency care visits', 'lower medication costs'.

This evaluation seeks to understand if targeted communication can effectively inform consumers about the availability of more affordable and generous health coverage options, thereby encouraging a shift towards plans that offer better value and accessibility.

ELIGIBILITY:
Inclusion Criteria:

* Households who qualify for automatic renewal of their Covered California health plan as of October 4.
* Households that were enrolled in Covered California on the subsidized application.

Exclusion Criteria:

Households that were no longer enrolled as of January 31, 2025. This includes people who chose to cancel their coverage in 2024 and those who were automatically disenrolled due to changes in eligibility during the open enrollment period.)

* Households that were included in the affordability crosswalk

  1. The affordability crosswalk is a Covered California process that moves eligible individuals with lower incomes to Silver CSR plans during renewal.
  2. This population includes members with incomes below 250% of the federal poverty level who were enrolled in Bronze plans and eligible for $0 premiums with Silver plans, members below 200% of the federal poverty level who were enrolled in Gold plans, and members below 150% of the federal poverty level who were enrolled in Platinum plans.
  3. Approximately 23,000 members are excluded from the experiment due to this restriction.
* Households with members enrolled with the carrier Valley Health Plan and Dental Health Services.

  1. This group was excluded due to changes in plan availability that necessitated a special notice.
  2. Approximately 30,000 members are excluded from this experiment due to this restriction.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600000 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment in an Enhanced CSR Plan | Up to 4 months
  A binary indicator for whether a consumer enrolled in an Enhanced CSR plan in 2025 open enrollment period.
Health care utilization outcomes among individuals enrolled in enhanced CSR plans in 2025. | 1 year
  Utilization will be assessed using binary indicators for various healthcare services, including primary care visits, emergency room visits, specialist visits, hospital admissions, and pharmacy claims. For each service type, the measure will reflect the number of visits or claims per 1,000 enrollees during the 2025 plan year.

SECONDARY OUTCOMES:
Consumer engagement: | Up to 4 months
  A binary indicator for consumers engagement including calls to service center, logins to user account, plan shopping on the website
Out-of-Pocket Health Care Spending | 1 year
  Measured as the total dollar amount spent by enrollees on out-of-pocket health care costs, including copayments, coinsurance, and deductibles, during the 2025 plan year.
Enrollment Tenure | 1 year
  Measured as the total duration of continuous enrollment in a health plan during the 2025 plan year, expressed in months. This outcome will assess whether receiving the educational flyer impacts the length of time enrollees remain covered.
Uninsured Status | 1 year
  A binary indicator identifying whether an individual has any uninsured months during the 2025 plan year, as determined by Franchise Tax Board (FTB) data.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kohn, Masters of Public Policy, Study Director — Covered California
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT07136233/Prot_SAP_000.pdf